CLINICAL TRIAL: NCT02290535
Title: Electrical Impedance Tomography of Lung in Child and Young Age
Acronym: EIT-Lunge
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 12-076; CIV-14-03-011942 (Other: Eudamed-Nr.)
Record Dates: First submitted 2014-09-19; First posted 2014-11-14 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Obstructive Lung Diseases
Keywords: obstructive pulmonary disease; children; teenager; EIT (Electrical Impedance Tomography)
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Children and Teenager of 5-18 years with obstructive pulmonary disease (asthma, cystic fibrosis, immotile-cilia-syndrome, obstructive bronchitis, obstructive pneumonia).
  Interventions: Procedure: patients
- Probands: Children and Teenager of 5-18 years without known obstructive pulmonary diseases
  Interventions: Procedure: probands

INTERVENTIONS:
Procedure: patients — The 16-electrode belt will be applied to patient's chest. Following vital signs will be recorded: respiratory rate at rest breathing, heart rate, transcutaneous oxygen saturation. Then impulse oscillometry (IOS) will be performed in a sitting position. After that, subjects with cooperation willingness will get a body plethysmography. A spirometry / forced breathing maneuvers will be performed. All patients will receive 2 strokes salbutamol inhaler for bronchospasmolysis. Please note that inhalation of salbutamol is not study related. It is used in the clinical routine to examine the reversibility of the bronchial obstruction in patients with obstructive lung disease in course of the lung function test. Ten minutes later measurements described above will be repeated.
  Groups: Patients
Procedure: probands — Probands will receive the same treatment as patients, but without bronchospasmolysis.
  Groups: Probands

SUMMARY:
The investigator will determine a compliance of two diagnostic techniques (EIT and Body plethysmography) in collective of children and teenagers with obstructive lung disease and a matched control group.

DETAILED DESCRIPTION:
The aim of the present study is verification of the correlation between EIT-derived data and following extracted parameters of the pulmonary function:

* forced expiratory volume in 1 second (FEV 1)
* forced vital capacity (FVC)
* relative forced expiratory volume in 1 second (FEV1/FVC)
* maximal expiratory flow (MEF 25)
* total lung capacity (TLC)
* resistance (Raw).

These findings could bring out new prospective opportunity for pulmonary function tests without cooperation.

Furthermore, the study aims to clarify whether EIT technique can be used for regional pulmonary function testing.

In addition, dynamic lung function parameter and static radiological techniques will be correlated with EIT.

ELIGIBILITY:
Inclusion Criteria:

* Patients: children and teenagers with obstructive pulmonary disease (asthma, cystic fibrosis, immotile-cilia-syndrome, obstructive brochitis, obstructive pneumonia).
* Probands: Children and Teenager of 5-18 years without known obstructive pulmonary diseases

Exclusion Criteria:

* active implants (ICD, CRT)
* metal in chest
* artificial heart valve
* children < 5 years
* pregnant and lactating females
* Persons, who are in relationship of dependence to the investigator / sponsor
* Persons, who are not able to understand and follow the instructions of the study personnel.
* Lack of signed informed consent (by legal guardian /proband)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients, who come to the consultation to the Department of Pediatric Pneumology, Children and Adolescent Medicine, University Hospital Aachen, will be recruited and divided into groups by age and diagnosis. Recriutment will be performed in accordance to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Robustness of change in electrical impedance based on the forced expiratory volume in 1 second (ΔZFEV01) | Baseline
  The robustness of ΔZFEV1.0 (= change in electrical impedance based on the FVC FEV1.0) and τ (= mechanical time constant τ which classifies the regional and global lung mechanics) and their clinical relevance will be investigated.

SECONDARY OUTCOMES:
Correlation between lung function parameters and extracted parameters of the EIT. | Baseline
  The present study aims to verify, whether a correlation between lung function parameters and extracted parameters of the EIT exists.
EIT as a diagnostic method for assessment of lung function | Baseline
  It will be examined, whether single EIT measurement can be used for assessment of the lung function.
Regional mechanical transmission behavior | Baseline
  Another secondary outcome is the local mechanical transmission behavior as an index of pulmonary status. By using the correlation between results gained from EIT and results from impulse oscillometry (IOS) differentiation between central and peripheral obstruction of respiratory tracts will be proved.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Lehmann, MD, Principal Investigator — Unversity Hospital Aachen
Locations (1):
- University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany